CLINICAL TRIAL: NCT00817076
Title: Evaluation of the Efficacy and Safety of Desloratadine Syrup in Childhood Atopic Dermatitis
Brief Title: Study of the Effectiveness and Safety of Desloratadine (Aerius) Syrup in Children With Allergic Skin Inflammation (P03475)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03475
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: desloratadine

INTERVENTIONS:
Drug: desloratadine — desloratadine syrup; 5.0 mL once daily for 28 days
  Other Names: Clarinex; Aerius; SCH 34117; descarboethoxyloratadine

SUMMARY:
The purpose of this study was to test the effectiveness and safety of desloratadine (Aerius) syrup in children with allergic skin inflammation. Patients took desloratadine syrup once a day for 28 days. Once a week, the doctor measured the patient's symptoms. This measurement is called SCORAD. The doctor also rated how much relief the patient got from treatment and recorded any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Children must be from >= 6 to < 12 years of age, of either sex and any race.
* Children's parent(s) or legal representative(s) must demonstrate their willingness to participate in the study and comply with its procedures by signing an informed consent.
* Children must be in general good health; i.e. they must be free of any clinically significant disease other than atopic dermatitis (AD) that would interfere with study evaluations.
* Children's parent(s) or legal representative(s) must understand and be able to adhere to the dosing and visit schedule, and agree to report concomitant medications and adverse events to the Investigator or designee.
* The diagnosis of AD will be performed according the Hanifin and Rajka criteria (Hanifin JM, Rajka G. Diagnostic features of atopic dermatitis. Acta Derm Venereol (Stockhr) 92 (suppl): 44-70, 1980): to be included in this study, children needed to manifest at least 3 major features and 3 minor features at visit 1 (day 1).
* Children must be clinically symptomatic with AD at visit 1 (day 1). Disease severity will be estimated using the SCORAD Index (European task force on atopic dermatitis. Severity scoring of atopic dermatitis: the SCORAD Index. Dermatology 186: 23-31, 1993), and child must have a SCORAD Index at least >= 35.

Exclusion Criteria:

* Children who have not observed the designated washout period for any of the prohibited medications.
* Children with bronchial asthma who require chronic use of inhaled or systemic corticosteroids.
* Children with a history of hypersensitivity to desloratadine, or any of its excipients.
* Children who have any current evidence of clinically significant hematopoietic, metabolic, cardiovascular, immunologic, neurologic, hematologic, gastrointestinal, hepatic, renal, psychiatric, or cerebrovascular, or any other disorder which, in the judgment of the Investigator, may interfere with the study evaluations or affect children safety.
* A known lack or response to H1-antihistamines.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2003-03; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Demonstration of the efficacy of desloratadine in relieving the total symptoms of atopic dermatitis through SCORAD Index | Baseline, Day 8, Day 15, and Day 29

SECONDARY OUTCOMES:
The percent of subjects who rate their response to desloratadine as either Complete, Marked, or Moderate Relief | Day 8, Day 15, and Day 29
Evaluate the number of adverse events during therapy | Day 8, Day 15, and Day 29